CLINICAL TRIAL: NCT02789267
Title: Nutrition and Quality of Life of Patients With Head and Neck Carcinoma After Radiotherapy
Acronym: NUQUE3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Rouen (Other); Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-A01684-45
Record Dates: First submitted 2016-03-17; First posted 2016-06-02 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2018-04

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Quality of Life; Dietary support
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Group of patients with standard of care: the nutritional support is conducted by physicians.
  No systematic dietary support
- Regular dietary support (Experimental): Group of patients will benefit from a systematic and regular dietary support. Patients will be followed by a dietitian 1 month and 3 month after radiotherapy in hospital. Then, dietitian will realize a telephon interview 2 and 5 months after radiotherapy
  Interventions: Other: Regular dietary support

INTERVENTIONS:
Other: Regular dietary support — Systematic and regular dietary support after radiotherapy
  Arms: Regular dietary support

SUMMARY:
Undernutrition in cancerology is frequent because it's present for thirty to fifty percent of the patients at the time of the diagnosis. According to the recommendations of the French Speaking Society of Clinical Nutrition and Metabolism (SFNEP) of November 2012, a five percent loss of weight compared to the previous weight increases the risk of toxicity of the chemotherapy and worsens the patient's quality of life.

The treatment of the tumors of the head and the neck comes along very often with a loss of weight (17.4 % after one year of radiotherapy according to the study of Larsson et al.) which varies with the chosen treatment, and shows a major risk at the patients whose therapeutic sequence involves a radiotherapy. The irradiation of the upper aerodigestive tract is source of aftereffects and late complications: xerostomia, oedemas of mucous membranes.

The xerostomia, connected to the damage of the salivary glands, is a frequent complaint of the patients. It reveals or even increases, a dysphagia. According to Woisard, six months after the end of treatments, forty percent of the patients suffer from a dysphagia.

All these complications limit quantitatively and qualitatively the food intake. The adaptation of the texture of the food is necessary by fifty four percent at three months of the end of treatments according to Logemann et al., and a few patients remain dependent on an long term enteral nutrition.

Beyond a change of the nutritional state, the feeding difficulties or even the absence of resumption of an oral feeding are responsible for a social isolation. The meal which lost its dimension of pleasure becomes a source of fear and obsession for the patient as well as for his relations, and this fact generates family tensions. The quality of life of the patient is heavily affected.

Ravasco showed in his study that the impact on the nutritional state of a nutritional care by dietary advices was more important as the prescription of oral nutritional supplements but based on a short period (the dietary intervention covered only the duration of the radiotherapy). But what would happen after the end of treatments? The investigators emit the hypothesis that a post-therapeutic systematic and regular dietary support has a positive impact on the prevention of the undernutrition among the patients affected by a first cancer of the upper aerodigestive tract whom therapeutic sequence involves a radiotherapy.

DETAILED DESCRIPTION:
The investigators propose a prospective randomized, open and multicentric study. This study has to include 224 patients affected by a head and neck cancer which therapeutic sequence involves a more or less made sensitized radiotherapy. The beginning of the inclusions is planned for May 2016, the end of inclusion 36 months later.

The nutritional state and quality of life will be evaluated 6 months after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with first head and neck cancer histologically proved
* treatment by radiotherapy
* no sign of recidive
* life expectancy 3-month-old superior
* OMS score < 3
* french speaking

Exclusion Criteria:

* other former cancer
* pregnant woman
* no oral feeding before radiotherapy
* uncontrolled infectious pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Patient's proportion presenting a decrease of 5% of their weight 6 months after the end of radiotherapy | 6 months
  the weight will measured by physician just after radiotherapy and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel BABIN, Pr, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No